CLINICAL TRIAL: NCT03913962
Title: Evaluation of Chronic Pathologies Impact and Their Treatments on Children and Teen Physical Fitness.
Brief Title: Health and Exercise Response in Children With Chronic and Auto-immune Pathologies
Acronym: HERCCULE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other); INSERM CIC 1405 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-409; 2018-A03247-48 (Other: 2018-A03247-48)
Record Dates: First submitted 2019-04-04; First posted 2019-04-12 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Juvenile Idiopathic Arthritis; Diabetes; Inflammatory Bowel Disease; Cancer Survivor; Anorexia Nervosa
Keywords: Paediatric; Auto-immunity; Treatment; Physical Activity
MeSH Terms: conditions — Arthritis, Juvenile; Diabetes Mellitus; Inflammatory Bowel Diseases; Anorexia Nervosa; Motor Activity | interventions — Calorimetry, Indirect

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): Patients with juvenile idiopathic arthritis, type 1 diabete mellitus, inflammatory bowel diseases, anorexia nervosa, cancer survivor
  Interventions: Other: indirect calorimetry
- Control (Active Comparator): healthy children sex- and age-matched
  Interventions: Other: indirect calorimetry

INTERVENTIONS:
Other: indirect calorimetry — Patients will be separated in different subgroups. Subgroups will be constituted according the disease status (i.e. active vs inactive) to assess the impact of the pathology on physical fitness and according to treatments to assess the effect of treatment on physical fitness.

SUMMARY:
The aim of the present project is to assess the effects of the chronic diseases and their associated treatments chronic paediatric diseases (CPD), to further understand their impact on physical fitness for public health perspectives. This is an innovative approach in the treatment of chronic paediatric diseases . This project should yield results that help improving treatments for children and adolescents with chronic paediatric diseases throughout physical activity as therapy, reduced pain, fatigue and inflammation, and improvement in physical fitness and life quality. The originality and novelty of this project is to combine architectural, functional and metabolic components of skeletal muscle to further understand the impact of chronic paediatric diseases as a function of treatment, disease activity and maturation status (prepubertal, pubertal or post pubertal).

This study will aim at assessing muscular function (force production capacity and fatigability) in specific or ecologic situations so as to get information about muscle functioning on isolated muscle group (here knee extensors) or during whole body exercise. Moreover, results arising from muscle architecture or quality will allow understanding the decrease in strength or endurance reported in the literature. The data collected will allow us to further understand the impact of the disease on structural, functional and metabolic parameters. Finally, the understanding of these alterations will provide information enabling to establish recommendations in physical activity (PA) to reduce or even counter the effect of the chronic inflammation and prevent at long-term overweight and cardiovascular risks.

The long-term objective is to contribute establishing recommendations or guidelines for prescribing physical activity during medical therapy. Values obtained in pathological children will be compared to those of control children matched for gender and maturation.

DETAILED DESCRIPTION:
Patients will be separated in different subgroups. Subgroups will be constituted according the disease status (active vs inactive) to assess the impact of the pathology on physical fitness and according to treatments to assess the effect of treatment on physical fitness.

Patients will perform physical tests to provide information about their physical fitness (body composition, metabolic flexibility, muscle strength and fatigue, bone mineral density), which will be compared to age- and gender-matched healthy controls. Patients will also complete blood tests to provide information about their inflammatory state to best understand physiological disorders and allow a better classification of the disease status.

1. Metabolic flexibility assessment

   After sitting quietly for 20 min, subjects will perform a graded exercise test to volitional fatigue on an electromagnetically braked cycle ergometer with continuous gas collection and heart rate monitoring. In all subjects, when the Respiratory Exchange Ratio will be ≥1.00, indicating zero fat oxidation, the work rate will be increased by the same increments at 1-min intervals until volitional fatigue. O2 consumption (VO2) peak will be considered maximal when the Respiratory Exchange Ratio will be ≥1.05 and the subject will achieve his age-predicted maximal heart rate [heart rate maximum: (220 - age)]. Indirect calorimetry, as will be used in this study, is the standard method to quantify substrate oxidation rates at rest and during exercise. O2 consumption (VO2) and CO2 production (VCO2) will be averaged over the final 1 min of each work rate, and the results of this test will be used to calculate fat oxidation over a wide range of exercise intensities for each subject with the equations:

   Lipids (mg.min-1) = 1.6946 x VO2 - 1.7012 x VCO2 and CHO (mg.min-1) = 4.585 VCO2 - 3.2255 VO2.
2. Muscle architecture Subjects will be lied on a massage table, muscle relaxed. Ultrasound will be used on vastus lateralis (VL), vastus medialis (VM) and rectus femoris (RF) to assess muscle architecture. The muscle belly will be measured according to Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) recommendations. Muscle thickness (the distance between superior and inferior aponeurosis) and fascicule angle (the angle formed by muscle fascicule and the inferior aponeurosis) will be measured for each muscle.
3. Muscle quality Subjects will sit on an adjustable seat. The right tight will be placed into the antenna of the peripheral quantitative tomography, so that the femoral condyles are aligned with the laser. An antero-posterior scout-view will be performed to detect junction between tibial tray and the femur, which matched with the starting position of the measurement. Then, a measure will be performed at 40% of the length between the greater trochanter and the mid-patella of the right leg. Muscle cross sectional area (CSA) and intramuscular adipose tissue (IMAT) will be assessed. The measurements will be performed by the same investigator to avoid any inter-individual bias.
4. Muscle function

   o Vertical jump height: Subjects will have to perform a series of vertical jumps. Subjects will perform two squat jumps (SJ) and two counter movements jumps (CMJ) using an OptoJump following standardised guidelines. For SJ, subjects will have to flex their knee at 90° with the hand on the hip to avoid any counter movements induced by the upper limbs. Subjects will have to maintain the position for 3-s. The guidelines for CMJ will be similar, but without short break between standing and flexing positions. For both exercises, subjects will have to jump as high as possible. Vertical jump height will be calculated according the formula where T is time flight duration and g the acceleration of 9.81 m.s-2 of gravity.

   o Maximal voluntary strength: Subjects will sit on an isokinetic dynamometer with a hip angle of 40° (0°= standing position). Upper body will be strapped on the chair back and subjects will have to grip the chair to avoid any counter-movements. Their right ankle will be strapped and connected to a force sensor. After a standardised warm up consisting of repeating isometric contractions at increasing intensities, patients will have to perform maximal voluntary isometric contractions (MVIC). MVIC will be performed at different randomized joint angles (29°, 66°, 76°, 87° and 103° [0° = full extension]) to determine the optimal angle producing maximal strength. Two measurements will be performed at each angle to check the reproducibility. A third trial will be performed if the difference between both measurements is higher than 5%. Subjects will be vigorously encouraged to produce maximal voluntary strength during isometric contractions. Root Mean Square (RMS) values will be calculated from the electromyographic (EMG) activity recorded on VL, VM and RF.
5. Muscle fatigue Muscle fatigue will be assessed with the same method as previously described. For this test, patients will have to maintain a force level corresponding to 50% MVIC to avoid any knee pain. The exercise will be stopped when subjects will be unable to maintain the force level more than 3-s despite vigorous encouragements. Time duration to task failure will be measured.
6. Bone micro-architecture Bone micro-architecture will be assessed through bone mineral density, trabecular and cortical density. This measurement will be performed in the same time that muscle quality assessment by pQCT. Patients will be placed in the same position. Two measurement will be done using pQCT at 20% and 40% of the tight. Micro-architectural parameters (trabecular and cortical density) will be calculated.
7. Body composition Body composition will be assessed by Dual-energy X-ray absorptiometry. Fat and fat-free mass, and bone density will be measured for the whole body and segments (arm, leg and trunk).
8. Biology Blood samples will be drawn once a year for patients and once for controls. Blood samples will allow to assess NFS (blood formul numeration), ionogramme, CRPus, VS, total bilirubin, ASAT, ALAT, GGT, PAL, glycaemia, total cholesterol -HDL-LDL, triglycerid, TSH, T4, adiponectin et leptin. Lipidomic, Cytokines and their receptors, calgranulins and MicroARNs will be also assessed thereafter.

ELIGIBILITY:
Inclusion Criteria:

* for patients:
* Aged between 6 and 18-year-old
* Male or female
* Presenting a chronic pathology / having a treatment which is known to alter muscle mass and function, metabolism and body composition
* Included in the active list of the hospital centre of Clermont-Ferrand
* Free and informed consent of the holders of parental authority and the patient
* Affiliated with the social security system for control:
* Aged between 6 and 18-year-old
* Male or female
* Free and informed consent of the holders of parental authority and the patient
* Affiliated with the social security system

Exclusion Criteria:

* for patients:
* Treatment by systemic corticoids (>1 week in the 30 days before test)
* Contraindication to sport practice
* Active infection for control:
* Contraindication to sport practice
* Chronic pathology susceptible to alter muscle mass and function, metabolism and body composition
* Treatment susceptible to alter metabolism
* Active infection

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal lipid oxidation rate during submaximal incremental exercise | at first test (at day 1)
  Percentage variation of the maximal strength rate during isometric contraction between pathological and healthy children

SECONDARY OUTCOMES:
Maximal strength during isometric contraction | at day 1
  Percentage variation of the maximal strength rate during isometric contraction between pathological and healthy children
Muscle architecture | At 6 months
  muscle cross sectional area (mm2) evaluated by peripheral Quantitative Computed Tomography (pQCT)
Body composition | At 6 months
  fat mass (g.cm²) evaluated by Dual-energy X-ray absorptiometry
Maximal muscular strength | At day 1
  maximal strength of knee extensors
Muscular fatigue | at 6 months
  Percentage variation of time to task failure duration during isometric contraction between pathological and healthy children.
Blood sample IL-17 | At day 1
  blood level of inflammation markers (IL-17)
Blood sample CRP | At day 1
  blood level of inflammation markers (CRP)
Blood sample IL-6 | At day 1
  blood level of inflammation markers (IL-6)
Blood sample TNF - a | At day 1
  blood level of inflammation markers (TNF - a)
Blood sample IL-10 | At day 1
  blood level of inflammation markers (IL-10a)
Blood sample INF | At day 1
  blood level of inflammation markers (INF)
Blood sample calprotectin | At day 1
  blood level of inflammation markers (calprotectin)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France